CLINICAL TRIAL: NCT00612027
Title: Trans GERD: Efficacy and Tolerability of Esomeprazol in Patients Under Ordinary Medical Care Conditions
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Dr Kai Richter, AstraZeneca Germany
Other Study IDs: 1312004011; German PMS trial no.9
Record Dates: First submitted 2008-01-29; First posted 2008-02-11 (Estimated); Last update posted 2008-02-11 (Estimated); Status verified 2008-01

CONDITIONS: Gastrointestinal Diseases
Keywords: gastrointestinal disorder; acid associated gastrointestinal symptoms.; esomeprazole therapy in patients with gastrointestinal disorders; patients with acid associated gastrointestinal symptoms
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: patients with gastrointestinal disorders and patients with acid associated gastrointestinal symptoms treated with esomeprazole.

SUMMARY:
Under daily routine conditions and without any intervention by the sponsor regarding the selection of subjects, diagnostic procedures, therapeutic decisions (medicinal and non- medicinal therapy, dose, duration, etc.), routine assessments, the participating physicians (i.e. general practitioners and internists) are asked to document relevant data related to esomeprazole therapy in patients with gastrointestinal disorders. Patients with acid associated gastrointestinal symptoms can be included.

ELIGIBILITY:
Inclusion Criteria:

* patients with gastrointestinal disorders and patients with acid associated gastrointestinal symptoms treated with esomeprazole.

Exclusion Criteria:

* limitiations; possible risks; warnings; contraindications mentioned in the SPC.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: general practitioners and internists
Sampling Method: Probability Sample
Enrollment: 29586 (Actual)
Dates: Start 2006-01; Primary Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
efficacy and tolerability of esomeprazole in patients who are treated by general practitioners and internists | proportion of treated subjects without any specific acid associated symptoms at the end of the study; change in intensity of specific acid associated symptoms; incidence of the occurrence of unknown, unexpected and/or rarely occurring adverse events AE.

SECONDARY OUTCOMES:
evaluation of a diagnosis tool | evaluation of the predictive value of a two items questionnaire on acid associated symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Kai Richter, MD, Study Chair — Medical Department AstraZeneca Germany